CLINICAL TRIAL: NCT05643586
Title: Effects of Ticagrelor Versus Prasugrel on Coronary Microcirculation in Patients Undergoing Elective Percutaneous Coronary Intervention: Results of the PROtecting MICROcirculation During Coronary Angioplasty (PROMICRO)-3 Randomised Study
Acronym: PROMICRO-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germano Di Sciascio (Other)
Collaborators: Cardiovascular Center Aalst, OLV Clinic, Aalst, Belgium (Unknown); Department of Advanced Biomedical Sciences, University of Naples Federico II, Italy (Unknown); CardioRISC, C-TRIC, Derry/Londonderry, Northern Ireland, UK (Unknown); University of Lausanne Hospitals (Other)
Responsible Party: Sponsor-Investigator, Germano Di Sciascio, Prof, Campus Bio-Medico University
Organization: Campus Bio-Medico University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2017/010
Record Dates: First submitted 2022-11-30; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Flow; Coronary Resistances; Platelet Reactivity
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to receive loading doses of either ticagrelor (180 mg) or prasugrel (60 mg) at least 12 hours before intervention. Assignment to one of the two treatments was determined by a computer-based randomization system.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization assignment for each patient was kept in a sealed envelope. At least 12 hours before PCI, a study nurse not involved in the procedure was responsible of opening the sealed envelope and administering study drugs according to treatment allocation. Both the patient and the catheterization laboratory team (operator and scrubbed nurse) were blinded to the assigned treatment. The PCI procedures were performed by standard technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prasugrel Group (Experimental): Patient treated with 60 mg prasugrel 12 hours before the procedure
  Interventions: Drug: Prasugrel
- Ticagrelor (Experimental): Patient treated with 180 mg ticagrelor 12 hours before the procedure
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Ticagrelor — Patient treated with 180 mg ticagrelor 12 hours before the procedure
  Other Names: Ticagrelor 180 mg
  Arms: Ticagrelor
Drug: Prasugrel — Patient treated with 60 mg prasugrel 12 hours before the procedure
  Other Names: Pasugrel 60 mg
  Arms: Prasugrel Group

SUMMARY:
Besides being at least as effective as prasugrel in inhibiting platelet aggregation, ticagrelor has been shown to have additional properties potentially affecting coronary microcirculation. We sought to compare the effects of ticagrelor and prasugrel on absolute coronary blood flow (Q) and microvascular resistance (R) in patients with stable coronary artery disease (CAD) undergoing elective percutaneous coronary intervention (PCI).

The PROMICRO-3 study shows that in patients with stable CAD undergoing PCI pre-treatment with a loading dose of ticagrelor compared with prasugrel improves post-procedural coronary flow and microvascular function and seems to reduce the related myocardial injury.

DETAILED DESCRIPTION:
Patient population We enrolled patients naïve to platelet P2Y12 receptor inhibitors with stable CAD referred to elective percutaneous coronary intervention (PCI) of an isolated, functionally significant (as confirmed by a fractional flow reserve [FFR] <0.80) stenosis located in the proximal two-thirds of a major coronary artery.

Study protocol Patients were randomly assigned to receive loading doses of either ticagrelor (180 mg) or prasugrel (60 mg) at least 12 hours before intervention. Assignment to one of the two treatments was determined by a computer-based randomization system and randomization assignment for each patient was kept in a sealed envelope. At least 12 hours before PCI (average 13.8±1.1), a study nurse not involved in the procedure was responsible of opening the sealed envelope and administering study drugs according to treatment allocation. Both the patient and the catheterization laboratory team (operator and scrubbed nurse) were blinded to the assigned treatment. The PCI procedures were performed by standard technique. In all cases, balloon pre-dilatation was performed before stent implantation.

Adjunctive medications All patients were administered a 500-mg loading dose of aspirin the day before the procedure. In the catheterization laboratory, all patients received a weight-adjusted intravenous heparin bolus (100 IU/kg) in order to maintain activated clotting time between 250 and 300 seconds. Patients randomized to the prasugrel group received clopidogrel 75 mg once daily as of the day after the PCI, whereas patients randomized to the ticagrelor group received a 600-mg loading dose the day after PCI, and a 75-mg maintenance dose as of the next day.8

Coronary physiology indexes Coronary physiology indexes were measured in each patient before and after PCI. Briefly, an intracoronary pressure/temperature sensor-tipped guide wire (PressureWire X, Abbott, IL) was advanced through the guiding catheter in the distal segment of the target coronary artery. A dedicated monorail catheter (RayFlow, Hexacath, Paris, France), allowing the infusion of saline through 4 outer side holes and the measurement of temperature by the guidewire through 2 inner side holes, was then advanced over the guidewire. The tip of the infusion catheter was placed in the first centimeter of the coronary artery, and the catheter was connected to an infusion pump (Medrad Stellant; Medrad Inc, Warrendale, PA), and saline at room temperature infused at a pre-specified flow rate (Qi, 20 mL/min for the left anterior descending [LAD] and left circumflex artery [LCx] and 15 mL/min for the right coronary artery [RCA]), resulting in a hyperaemic state similar to that produced by adenosine. The temperature of the saline/blood mixture (T) and the distal coronary pressure (Pd) were measured after achieving a steady state. Aortic pressure (Pa) was measured through the guiding catheter. Fractional flow reserve (FFR) was calculated as Pd/Pa during hyperaemia. The temperature of the infused saline (Ti) was measured after pulling the temperature sensor of the guidewire back into the infusion catheter. Pressure tracings and temperatures were simultaneously analysed by a dedicated console equipped with software that automatically calculates physiology indexes (Coroventis Coroflow, Uppsala, Sweden). Q was calculated as 1.08 x (Ti/T) x Qi, and expressed in ml/min. Following the Ohm's law, R was calculated as Pd/Q, and expressed as mm Hg/L/min, or Wood units.

Platelet function analysis Platelet reactivity was measured before study drug assignment and at the time of PCI using the VerifyNow P2Y12 assay (Accumetrics, San Diego, California). The VerifyNow P2Y12 assay is a validated optical turbidimetric point-of-care assay specifically assessing the effects of P2Y12 receptor inhibitors:12 the results are reported as P2Y12 reaction units (PRU), and the lower the PRU value, the higher the platelet aggregation inhibition.

Peri-procedural myocardial injury High sensitivity Troponin I (hs-TnI; Roche Diagnostics, Mannheim, Germany) was determined in blood samples taken before, 8 and 24 hours after the intervention. Peak post-PCI hs-TnI levels were considered for the analysis.

Statistical analysis At the time the study was conceived, no published data were available on this topic. However, an estimate of Q values was assumed from preliminary data collected at our Institution.10 Expecting a 20% reduction in post-PCI R with ticagrelor compared with prasugrel (320±75 vs 400±85 mmHg/l/min), a total of at least 23 patients per group were needed to achieve 90% power at a 2-sided alpha of 0.05 to detect the anticipated difference. Therefore, we aimed at enrolling a total of 50 patients (25 per group). Continuous variables are expressed as mean ± SD or as median [25th, 75th percentile], as appropriate. Categorical variables are reported as frequencies and percentages. Normal distribution was tested with the Shapiro-Wilk W test. Comparisons between continuous variables were performed using the Student t test or Mann-Whitney test. These tests were corrected for repeated measures where appropriate. Repeated measures 2-way analysis of variance (ANOVA) was used to assess the effect interaction between treatment and time on continuous variables. Comparisons between categorical variables were evaluated using the Fisher exact test or the Pearson chi-square test, as appropriate. Correlations between continuous variables were assessed using the Spearman correlation test. Statistical analysis was performed using STATA/IC 14 (STATA Corp., College Station, Texas) and p values <0.05 (two tailed) were considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Paitents with stable CAD referred to elective percutaneous coronary intervention (PCI) of an isolated, functionally significant (as confirmed by a fractional flow reserve [FFR] <0.80) stenosis located in the proximal two-thirds of a major coronary artery

Exclusion Criteria:

* age <18 years or ≥75 years, body weight <60 kg, previous transient ischemic attack (TIA) or stroke, acute coronary syndromes, administration of glycoprotein IIb/IIIa inhibitors, platelet count <70x109/l, high bleeding risk (active internal bleeding, history of haemorrhagic stroke, intracranial neoplasm, arteriovenous malformation or aneurysm, ischemic stroke in the previous 3 months), coronary bypass graft surgery in the previous 3 months, severe chronic renal failure (serum creatinine ≥2 mg/dl), previous myocardial infarction, left ventricular ejection fraction less than 50%, left ventricle wall-motion abnormalities, left ventricular hypertrophy, chronic total occlusion, lesions with extensive calcifications requiring rotational atherectomy, in-stent restenosis, bifurcation lesions with side branch diameter of more than 2 mm, ostial lesion, and contraindications to adenosine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-04-14 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Post PCI coronary flow | Immediately after the procedure
  Post PCI flow measured according to continous termodiluition
Post PCI coronary resistance | Immediately after the procedure
  Post PCI coronary resistance measured according to continous termodiluition

SECONDARY OUTCOMES:
Periprocedural myocardial injury | 8 and 24 hours following the procedure
  cTn elevation following PCI

CONTACTS AND LOCATIONS:
Locations (1):
- Aalst cardiovascular center, Aalst, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Available following reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Mangiacapra F, Peace AJ, Di Serafino L, Pyxaras SA, Bartunek J, Wyffels E, Heyndrickx GR, Wijns W, De Bruyne B, Barbato E. Intracoronary EnalaPrilat to Reduce MICROvascular Damage During Percutaneous Coronary Intervention (ProMicro) study. J Am Coll Cardiol. 2013 Feb 12;61(6):615-21. doi: 10.1016/j.jacc.2012.11.025. Epub 2013 Jan 2. PMID 23290547
- [Background] Mangiacapra F, Di Gioia G, Pellicano M, Di Serafino L, Bressi E, Peace AJ, Bartunek J, Wijns W, De Bruyne B, Barbato E. Effects of Prasugrel Versus Clopidogrel on Coronary Microvascular Function in Patients Undergoing Elective PCI. J Am Coll Cardiol. 2016 Jul 12;68(2):235-7. doi: 10.1016/j.jacc.2016.04.039. No abstract available. PMID 27386781
- [Background] Cattaneo M, Schulz R, Nylander S. Adenosine-mediated effects of ticagrelor: evidence and potential clinical relevance. J Am Coll Cardiol. 2014 Jun 17;63(23):2503-2509. doi: 10.1016/j.jacc.2014.03.031. Epub 2014 Apr 23. PMID 24768873
- [Background] Jaffe R, Dick A, Strauss BH. Prevention and treatment of microvascular obstruction-related myocardial injury and coronary no-reflow following percutaneous coronary intervention: a systematic approach. JACC Cardiovasc Interv. 2010 Jul;3(7):695-704. doi: 10.1016/j.jcin.2010.05.004. PMID 20650430
- [Background] Xaplanteris P, Fournier S, Keulards DCJ, Adjedj J, Ciccarelli G, Milkas A, Pellicano M, Van't Veer M, Barbato E, Pijls NHJ, De Bruyne B. Catheter-Based Measurements of Absolute Coronary Blood Flow and Microvascular Resistance: Feasibility, Safety, and Reproducibility in Humans. Circ Cardiovasc Interv. 2018 Mar;11(3):e006194. doi: 10.1161/CIRCINTERVENTIONS.117.006194. PMID 29870386
- [Background] Gallinoro E, Candreva A, Colaiori I, Kodeboina M, Fournier S, Nelis O, Di Gioia G, Sonck J, van 't Veer M, Pijls NHJ, Collet C, De Bruyne B. Thermodilution-derived volumetric resting coronary blood flow measurement in humans. EuroIntervention. 2021 Oct 1;17(8):e672-e679. doi: 10.4244/EIJ-D-20-01092. PMID 33528358
- [Background] Mangiacapra F, Barbato E, Patti G, Gatto L, Vizzi V, Ricottini E, D'Ambrosio A, Wijns W, Di Sciascio G. Point-of-care assessment of platelet reactivity after clopidogrel to predict myonecrosis in patients undergoing percutaneous coronary intervention. JACC Cardiovasc Interv. 2010 Mar;3(3):318-23. doi: 10.1016/j.jcin.2009.12.012. PMID 20298992
- [Derived] Mangiacapra F, Colaiori I, Di Gioia G, Pellicano M, Heyse A, Paolucci L, Peace A, Bartunek J, de Bruyne B, Barbato E. Effects of ticagrelor and prasugrel on coronary microcirculation in elective percutaneous coronary intervention. Heart. 2023 Dec 20;110(2):115-121. doi: 10.1136/heartjnl-2022-321868. PMID 37316163